CLINICAL TRIAL: NCT04331548
Title: Study Of Endobronchial Ultrasound Transbronchial Needle Aspiration (EBUS-TBNA) Cytology Of Enlarged Mediastinal & Hilar Lymph Nodes Detected In Interstitial Lung Disease
Brief Title: Endobronchial Ultrasound Transbronchial Needle Aspiration Of Enlarged Mediastinal In Interstitial Lung Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Liran Levy, Principal Investigator, Sheba Medical Center
Other Study IDs: SHEBA-20-7006-20-SMC-LL-CTIL
Record Dates: First submitted 2020-03-22; First posted 2020-04-02 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the findings of mediastinal/hilar LN sampling by EBUS-TBNA in patients with non-sarcoidosis interstitial lung disease ( ILD) who demonstrate LN enlargement on chest imaging. Patients with non-sarcoidosis ILD referred for bronchoscopy will undergo LN sampling by EBUS-TBNA. Cytology results will be recorded along with clinico-radiologic features, BAL findings, histology and final ILD diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. non-sarcoidosis ILD (low probably of sarcoidosis based on radiology),
2. referred for bronchoscopy (BAL, TBLB or TBCB) in the Interventional Pulmonology Unit at Sheba Medical Center
3. Patients with LN enlargement ≥1 cm in short diameter at stations 2, 4, 7, 10 or 11 (LN stations accessible to EBUS-TBNA)

Exclusion Criteria:

1. known ILD
2. ILD with no indication to bronchoscopy
3. contraindication to bronchoscopy .

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients referred for bronchoscopy (BAL, TBLB or TBCB) in the Interventional Pulmonology Unit at Sheba Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-05-30 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
assessing the findings of mediastinal/hilar LN sampling by EBUS-TBNA in patients with non-sarcoidosis ILD who demonstrate LN enlargement on chest imaging. | during the procedure/surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel